CLINICAL TRIAL: NCT00005242
Title: Childhood Passive Smoking: Cohort Study of Cardiac Risk
Status: Completed | Type: Observational
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1123; R29HL038878 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2016-02

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Lung Diseases; Coronary Arteriosclerosis
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Lung Diseases; Coronary Artery Disease

SUMMARY:
To determine the effects of long-term exposure to passive smoking on the cardiovascular and oxygen transport systems in pre-adolescent twins.

DETAILED DESCRIPTION:
BACKGROUND:

The adverse health effects of actively inhaled cigarette smoke include impaired pulmonary function, increased coronary and cerebrovascular disease, chronic pulmonary disease, and cancer. Infants and young children of smoking parents are at increased risk for lower respiratory tract infections and small airways disease than are children of non-smoking parents. What is less clear is how the oxygen transport system of the growing child is affected by the long-term exposure to and passive inhalation of cigarette smoke and if this exposure represents a risk for the subsequent development of atherosclerotic heart disease.

DESIGN NARRATIVE:

A sample of 300 pre-adolescent twin pairs was recruited from an established population-based twin study. The three cohorts of twins and their parents were initially evaluated in a cross-sectional study and then followed longitudinally for up to three years. In the initial testing cycle the following data were collected: genotype; general health; anthropometric measures; resting and exercise noninvasive evaluation of hemodynamic parameters including blood pressure, heart rate, cardiac output, left ventricular mass, and oxygen consumption; hematocrit and blood levels of 2,3-DPG, cotinine, thiocyanate, and erythropoietin; spirometric and pulmonary flow data; lipid levels. There were three follow-up exams. The availability of repeated measures of oxygen delivery and its determinants in twins and their parents permitted both a unique analysis of genetic and environmental factors during the process of developmental change and measurements of the risks of accelerated atherosclerotic/ischemic heart disease and of the development of reactive airway disease.

The following hypotheses were tested: genetic factors accounted for a significant proportion of the variation in the hematologic and cardiovascular determinants of systemic oxygen delivery; adaptive responses of the oxygen delivery system differed in the same individual before and after puberty; passive smoking in children was an incremental risk factor for the development of accelerated atherosclerotic/ischemic cardiovascular disease; passive smoking in children was a contributing factor in the development of reactive airway disease.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1989-04; Study Completion 1994-06

REFERENCES:
- [Background] Moskowitz WB, Mosteller M, Schieken RM, Bossano R, Hewitt JK, Bodurtha JN, Segrest JP. Lipoprotein and oxygen transport alterations in passive smoking preadolescent children. The MCV Twin Study. Circulation. 1990 Feb;81(2):586-92. doi: 10.1161/01.cir.81.2.586. PMID 2297864
- [Background] Schieken RM, Mosteller M, Goble MM, Moskowitz WB, Hewitt JK, Eaves LJ, Nance WE. Multivariate genetic analysis of blood pressure and body size. The Medical College of Virginia Twin Study. Circulation. 1992 Dec;86(6):1780-8. doi: 10.1161/01.cir.86.6.1780. PMID 1451250
- [Background] Goble MM, Mosteller M, Moskowitz WB, Schieken RM. Sex differences in the determinants of left ventricular mass in childhood. The Medical College of Virginia Twin Study. Circulation. 1992 May;85(5):1661-5. doi: 10.1161/01.cir.85.5.1661. PMID 1572024
- [Background] Newkumet KM, Goble MM, Young RB, Kaplowitz PB, Schieken RM. Altered blood pressure reactivity in adolescent diabetics. Pediatrics. 1994 Apr;93(4):616-21. PMID 8134217
- [Background] Moskowitz WB, Mosteller M, Hewitt JK, Eaves LJ, Nance WE, Schieken RM. Univariate genetic analysis of oxygen transport regulation in children: the Medical College of Virginia Twin Study. Pediatr Res. 1993 Jun;33(6):645-8. doi: 10.1203/00006450-199306000-00022. PMID 8378126